CLINICAL TRIAL: NCT04418375
Title: Identification of Markers Associated With the Risk of COVID-19 Infection and Symptomatic COVID+ Versus Asymptomatic COVID+ Status Through the Establishment of a Biological Collection During Serological Screening in APHP Professionals
Brief Title: Establishment of a Biological Collection During COVID-19 Serological Screening in APHP Professionals (COVID-HOP)
Acronym: COVID-HOP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Université de Paris (Unknown); Fondation Hôpitaux de Paris-Hôpitaux de France (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP200609; APHP200609 (Other: Assistance Publique - Hôpitaux de Paris); 2020-A01364-35 (Other: IDRCB)
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Serology,; Immunity; Hospital staff; Biobank
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum (12 mL), Plasma (EDTA 12 mL, citrate 7 mL), Peripheral blood mononucleated cells (PBMC), DNA, RNA, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the COVID-HOP study is to identify biological and non-biological markers associated to: a positive or negative serology anti SRAS-Cov-2; a positive serology and having presented symptoms or, on the contrary, not having had symptoms; the persistence of immunity or the loss of this immunity over time; the protective nature of the presence of anti SRAS-Cov-2 antibodies.

To answer these questions, a biological collection (serum, plasma, DNA, RNA, mono-nucleated cells and urine) and a collection of detailed clinical data during the serological screening for SARS-CoV-2 of hospital agents (medical and non-medical staff) of the Assistance Publique Hôpitaux de Paris (Paris, France) will be carried out. 4000 professionals in 5 hospitals will be included. As part of the research, the anti SRAS-CoV-2 serology will be monitored 6 months and 12 months after the initial serology. Numerous studies will be carried out from this biological collection and from the database to answer the primary and secondary endpoints.

DETAILED DESCRIPTION:
To answer the questions raised in the primary and secondary endpoints, a biological collection (serum, plasma, DNA, RNA, mono-nucleated cells and urine) and a collection of detailed data by the mean of a questionnaire (demographic, clinical, lifestyle, professional exposure to the virus, COVID-19 infection with detailed symptoms and complications) during the serological screening for SARS-CoV-2 of hospital agents (medical and non-medical staff) of the Assistance Publique Hôpitaux de Paris (Paris, France) will be carried out. 4000 professionals in 5 hospitals of the Assistance Publique Hôpitaux de Paris. As part of the research, the anti SRAS-CoV-2 serology will be monitored 6 months (M6) and 12 months (M12) after the initial serology and a brief questionnaire (update regarding treatments, co-morbidities, and COVID-19 infection) will be fulfilled at these two time points. Of note, if the inclusion could not be performed during the initial serological screening, the professional will be recalled to be included at M6.

Statistical analysis: The analysis of the determinants independently associated with symptomatic COVID + status will be carried out by uni- and multivariate logistic regression. The internal validation will be carried out by methods of draw with discount (bootstrap). The performance of the model will include calibration (graphical method) and discrimination (AUC). The biomarker study will include the study of the association with COVID + symptomatic versus asymptomatic status by univariate then multivariate analyzes (logistic regression) including clinical variables. The additional value of biomarkers will be studied by comparing the discriminating power of clinical models with and without the new biomarker. Finally, the study of the heterogeneity of COVID + symptomatic and asymptomatic patients will be carried out by an unsupervised analysis of Machine Learning known as archetypes.

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff (medical and non-medical)
* Age greater than or equal to 18 years
* Benefiting from or having benefited 6 months ago from carrying out a SARS-CoV-2 serology by venous sampling on a APHP site as part of monitoring by a screening center
* Having been informed about the study and having given their informed consent to participate in the study
* Beneficiary or entitled to a social security scheme

Exclusion Criteria:

* Refusal to participate in the study
* Previously known anemia with hemoglobin <10 g / dL
* Subject already included in a cohort study with biological collection COVID-19
* Exclusion period for subjects included or having been included in a COVID-19 interventional study (prophylactic or curative) or other clinical study
* Subject who received blinded treatment for SARS-Cov-2 in a clinical study
* Recent COVID-19 compatible infection with D0 of symptoms less than 4 weeks before collection
* Subject subject to a judicial protection measure
* Subject under guardianship or curatorship
* Subject under state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital staff agent (medical and non medical) from the "Assistance Publique Hôpitaux de Paris" undergoing a serology to depict IgG anti SRAS-Cov-2 antibodies in a screening center from the "Assistance Publique Hôpitaux de Paris" .
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Identification of markers associated with asymptomatic COVID + status (results of the serological test) versus symptomatic COVID + status through a questionnaire (medical history, work environment, lifestyle) and a biological collection | 12 months

SECONDARY OUTCOMES:
Identification of markers associated with a positive or a negative serology through a questionnaire (medical history, work environment, lifestyle) and a biological collection | 12 months
Description of the serological status according to the professional risk of exposure to the virus | 12 months
  The level of risk of occupational exposure to SARS-CoV-2 will be described in detailed (type of activity during the COVID-19 pandemic, type of protection during this activity...)
Description of the clinical manifestations of COVID-19 infection in hospital professionals | 12 months
  All the potential clinical signs of a COVID-19 infection and its complication will be recorded
Identification of risk factors associated with the loss of anti SARS-CoV-2 immunity through a questionnaire (medical history, work environment, lifestyle) and a biological collection | 12 months
Identification of markers associated with symptomatic COVID-19 infection during follow-up despite the presence of anti SARS-CoV-2 antibodies through a questionnaire (medical history, work environment, lifestyle) and a biological collection | 12 months
Correlation between the serology result and the PCR result (swabs) for people who have been tested as part of routine care. | 12 months
  Correlation between the serology result and the PCR result (swabs) for people who have been tested by PCR as part of routine care.
Identification of potential therapeutic targets to avoid developing a symptomatic form | Through study completion, an average of 2 years
  purpose of potential ancillary studies using the biological collection
Identification of potential therapeutic targets to promote the maintenance of an anti SARS-CoV2 protective immunity | Through study completion, an average of 2 years
  purpose of potential ancillary studies using the biological collection
Creation of COVIDneg and COVID + asymptomatic control groups for other COVID-19 biological collections. | Through study completion, an average of 2 years
  purpose of the biological collection that will include people with a negative SRAS-CoV-2 serology and asymptomatic people with a positive SRAS-CoV-2 serology

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Dr DEMORY, PhD, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou, Paris; Solen Dr KERNEIS, PhD, Principal Investigator — AP-HP, Hôpital Cochin, Paris; Martine Dr LOUET, PhD, Principal Investigator — AP-HP, Hôpital la Pitié Salpêtrière, Paris; Bénédicte Dr SAWICKI, PhD, Principal Investigator — AP-HP, Hôpital Bichat, Paris; Véronique Dr MAHE, PhD, Principal Investigator — AP-HP, Hôpital Lariboisière, Paris
Locations (1):
- HEGP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: from february 2021 for the primary outcome and as long as samples will be available in the biological collection.
Access Criteria: Ancillary studies willing to use the biological collection and/or dataset of the COVID-HOP study will be submitted to the scientific board of COVID-HOP for evaluation.
  Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization

REFERENCES:
- [Derived] Smadja DM, Roux de Bezieux J, Peronino C, Jilet L, Ivak P, Pya Y, Philippe A, Latremouille C, Gustafsson F, Ramjankhan FZ, Roussel JC, Courbebaisse M, Parfait B, Lebeaux D, Friedlander G, Vincentelli A, Flecher E, Gaussem P, Jansen P, Netuka I. Understanding Platelet Activation in the Aeson Bioprosthetic Total Artificial Heart: Insights From Aspirin Treatment and Outcomes. ASAIO J. 2025 Sep 1;71(9):701-710. doi: 10.1097/MAT.0000000000002403. Epub 2025 Feb 28. PMID 40019017